CLINICAL TRIAL: NCT04009889
Title: Double Blind,Randomized, Controlled Trial on Impact of Oral Probiotic Blend ( Lactobacillus Rhamnosus GG, L. Crispatus LBV88, L. Rhamnosus LBV96, L.Jensenii LBV116 and L. Gasseri LBV150 ) on Pregnancy Outcome
Brief Title: Impact of Oral Probiotic Blend on Pregnancy Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i-Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSO-PregO-2018
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
MeSH Terms: interventions — calcium D-pantothenate, L-cysteine drug combination; stearic acid; Silicon Dioxide

STUDY DESIGN:
Intervention Model Description: N=162 pregnant women were randomly assigned to one of the 2 interventions: verum (Lactobacilli) or placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- verum (Active Comparator): probiotic bland with 5 different lactobacilli
  Interventions: Dietary Supplement: capsule containing a probiotic blend of 5 different Lactobacilli
- placebo (Placebo Comparator): Microcrystalline Cellulose, Magnesium Stearate, Silicon Dioxide, but no probiotics.
  Interventions: Other: capsule containing Microcrystalline Cellulose, Magnesium Stearate, Silicon Dioxide, but no probiotics.

INTERVENTIONS:
Dietary Supplement: capsule containing a probiotic blend of 5 different Lactobacilli — n=81 women (verum) starts before end of pregnancy week 14 with consumption of 1 capsule daily until delivery.
  Other Names: verum
  Arms: verum
Other: capsule containing Microcrystalline Cellulose, Magnesium Stearate, Silicon Dioxide, but no probiotics. — n=81 women (placebo) starts before end of pregnancy week 14 with consumption of 1 capsule daily until delivery.
  Other Names: placebo
  Arms: placebo

SUMMARY:
The aim of this study is, to investigate the effect of oral intake of Lactobacillus rhamnosus GG (ATCC 53103), Lactobacillus crispatus Lbv88, Lactobacillus rhamnosus Lbv96, Lactobacillus jensenii Lbv116 Lactobacillus gasseri Lbv150 on outcomes of pregnancy and microbiota and their interrelation.

DETAILED DESCRIPTION:
Pregnant women aged > 18 years in the < 14th week of pregnancy willing to consume the study product once daily starting the day after V1 until delivery, complying with inclusion and exclusion criteria will be enrolled in the study.

After enrollement subjects will be randomly and evenly assigned to one of the two test groups verum and placebo.

The study population will be recruited in a screening examination ( G1 ) by gynaecologists from Kiel area.

Primary target parameter of the study :

HOMA-IRa value in week 24-28 (V2), which is based on glucose and insulin measures during the second oral glucose tolerance test (OGTT)

Secondary target parameters :

HOMA-IR value in week 36-40 , Alteration (V2 - V1) Δ HOMA-IR, Alteration (V2 - V1) Δ QUICKI

ELIGIBILITY:
Inclusion Criteria:

* pregnant women aged > 18 years in the < 14 week of pregnancy
* willing to consume the study product during pregnancy ( V1 to delivery)
* willingness to abstain from probiotic food and supplements containing probiotics
* written informed consent

Exclusion Criteria: Any of the following is regarded as a criterion for exclusion from enrollment in the study:

1. Subjects currently enrolled in another clinical study
2. Subjects having finished another clinical study within the last 4 weeks before inclusion
3. Diabetes mellitus
4. Acute metabolic disorder interfering with glucose metabolism
5. Known cancer < 5y ago
6. Any ano-rectal infection, disease, surgery in the medical history or current which may have impact on microbiota
7. Anus praeter
8. Hypersensitivity, allergy or idiosyncratic reaction to any component of the test product
9. Any disease or condition which might significantly compromise the hematopoietic, renal, endocrine, pulmonary, hepatic, gastrointestinal, cardiovascular, immunological, central nervous, dermatological or any other body system
10. History of active hepatitis B and C
11. History of HIV infection
12. Regular medical treatment including OTC, which may have impact on the study aims (e.g. probiotics, antibiotic drugs, laxatives etc.)
13. Major cognitive or psychiatric disorders
14. Present drug abuse or alcoholism, reformed alcoholic Legal incapacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women aged > 18 years in the < 14 week of pregnancy
Enrollment: 170 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
HOMA-IR value in week 24-28 | measurement between 24-28 week of pregnancy
  HOMA -IR is the product of insulin x glucose and describes the level of insulin resistance
HOMA-IR value in week 36-40 | measurement between 36-40 week of pregnancy
  HOMA -IR is the product of insulin x glucose and describes the level of insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Laue, MD, Principal Investigator — Clinical Research Center Kiel GmbH, Germany
Locations (1):
- Clinical Research Center Kiel GmbH, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Davidson SJ, Barrett HL, Price SA, Callaway LK, Dekker Nitert M. Probiotics for preventing gestational diabetes. Cochrane Database Syst Rev. 2021 Apr 19;4(4):CD009951. doi: 10.1002/14651858.CD009951.pub3. PMID 33870484